CLINICAL TRIAL: NCT04184609
Title: Mechanisms for Dyspnea on Exertion in Children With Obesity and Asthma: Distinct Physiological Phenotypes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding ran out before participants were enrolled.
Sponsor: Ohio State University (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Dharini Bhammar, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1481566
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Asthma in Children; Dyspnea; Asthmatic; Obesity, Childhood
Keywords: Pediatric; Breathlessness; Ventilatory Constraints; Exercise
MeSH Terms: conditions — Dyspnea; Asthma; Pediatric Obesity; Motor Activity | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: 2 repeated measures (within factor): Control and Albuterol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise test (Experimental): All participants will undergo a moderate-intensity exercise test under three conditions in a repeated measures study design:
  1. Control
  2. Albuterol
  Interventions: Other: Control; Drug: Albuterol

INTERVENTIONS:
Other: Control — In this condition, the participants will not receive any medications or drugs before exercise
  Other Names: No-treatment
Drug: Albuterol — 180 mcg of Albuterol will be administered before exercise
  Other Names: Ventolin

SUMMARY:
The overall objective of this study is to better understand the respiratory mechanisms provoking dyspnea on exertion in obese asthmatic children.

DETAILED DESCRIPTION:
Obesity and asthma are the most common diseases of childhood, causing activity limitation and impaired quality of life. Most obese asthmatic children report dyspnea on exertion (DOE) as their primary asthma symptom. Fear of dyspnea promotes sedentariness and reduces exercise capacity and quality of life. DOE in asthmatic children is typically attributed to bronchoconstriction but it is also possible that obesity is an equal or even major contributor to dyspnea. Excess chest and abdominal weight in obese children results in low lung volumes, which increases the risk of mechanical ventilatory constraints such as expiratory flow limitation, dynamic hyperinflation, and airway closure, all of which can provoke DOE. Unnecessary use of corticosteroids and other asthmatic medication in obese asthmatic children cannot treat obesity-specific mechanical ventilatory constraints and could have unintended deleterious effects. Therefore, there is an urgent need to better understand the mechanisms involved in DOE to provide evidence-based symptom management for obese asthmatic children that will promote regular physical activity and lessen DOE.

The overall objective of this study is to better understand the respiratory mechanisms provoking DOE in obese asthmatic children. The investigators hypothesize that low lung volume breathing in obesity leads to mechanical ventilatory constraints in the presence or absence of bronchoconstriction during exercise. Whereas DOE attributable to bronchoconstriction should respond to bronchodilators, DOE attributable to obesity-specific mechanical ventilatory constraints will not respond to bronchodilators. A comprehensive physiological pulmonary function and exercise-testing based approach will be used to identify 9-17-year-old obese asthmatic children who do and do not bronchoconstrict during exercise. The presence/absence of bronchoconstriction will be determined by a comprehensive measure of exercise-induced central and peripheral airway reactivity using spirometry and impulse oscillometry (i.e., greater than or equal to 10% reduction in forced expiratory volume in 1s, FEV1, or greater than or equal to 40% increase in peripheral airway resistance, R5-20, will be indicative of bronchoconstriction). The investigators will also determine the mechanisms by which bronchodilators like albuterol affect bronchoconstriction amd mechanical ventilatory constraints in asthmatic children with obesity.

ELIGIBILITY:
General inclusion criteria:

* Age range: 9-17 years of age
* Participants with physician diagnosed asthma will be recruited for this study.

  * Objectively Confirmed Asthma Diagnosis: Asthma diagnosis will be confirmed objectively using spirometry (FEV1 < 80% predicted or FEV1/FVC < lower limit of normal), bronchodilator reversibility testing (post-bronchodilator improvement of ≥ 12% and 200mL in FEV1 or FVC; or a decrease in lung hyperinflation of at least 150 mL; ATS guidelines on lung function test interpretation). Patients in whom asthma cannot be confirmed objectively will be excluded from the study.
* Experience dyspnea on exertion as assessed by answering "yes" to one of the following two questions on the screening questionnaire: 1) Do you get short of breath with exertion? 2) Do you feel that your asthma is limiting you from participating in exercise?
* Ability to communicate in English

Body mass index criteria (BMI): We will study asthmatic children with obesity based on their BMI percentile:

• Obese: BMI ≥95th percentile and less than 170% of the 95th BMI percentile based on norms from the CDC

Exclusion criteria:

Criteria for pulmonary function: We will exclude asthmatic children with:

* Severe asthma: Forced expiratory volume in 1s (FEV1) < 50% predicted
* Restrictive pulmonary disease: Forced vital capacity (FVC) and total lung capacity (TLC) < 80% predicted
* Diffusion limitation: Diffusing capacity relative to alveolar volume (DLCO/VA) < 80% predicted

Daily activity levels: Children participating in regular vigorous conditioning exercise such as running, jogging, aerobics, cycling, or swimming for ≥60min/session and ≥five times per week will be excluded to ensure similarity in physical activity levels between subjects and to avoid enrolling a potential high-fit, extremely active child. Children who participate in daily, unorganized physical activity (i.e., majority of children), will not be excluded. Children who are sedentary or only participate in school physical education classes will not be excluded.

The following exclusion criteria will be used in this study:

* History of oral steroid medications for 4 weeks prior to enrollment
* History of being admitted to an intensive care unit or being intubated because of their asthma in the past five years
* History of allergy or hypersensitivity to albuterol
* On long acting muscarinic antagonists (LAMA)
* History of vocal cord dysfunction
* History of obesity hypoventilation syndrome
* History of untreated sleep apnea
* History of heart disease, metabolic disease, or renal disease that, in the opinion of the PI (or co-I's), would increase the risks of exercise testing or alter the physiological responses to exercise
* History of significant mental illness that in the opinion of the PI (or co-I's) would interfere with study participation or increase risks to the participant
* History of musculoskeletal abnormality that would preclude cycling exercise
* Pregnant or become pregnant during their participation in the study
* History of other significant illnesses that, in the opinion of the PI (or co-I's), either increase risks of participation or alter the physiological responses to exercise
* Inability to successfully complete pulmonary function or exercise testing measurements or difficulty with following instructions during testing
* Inability to tolerate testing procedures or complications related to testing
* If a participant develops hypoxemia or meets indications for terminating exercise, the exercise test will be terminated, and the participant will be referred for further evaluation In general, all participants will be encouraged to follow up with their asthma care provider or pediatrician for any health concerns that are discovered during their participation.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Expiratory flow limitation | up to 2 hours during the intervention (exercise)
  Units: % of tidal volume, measured as overlap between exercise tidal flow volume loop and maximal expiratory flow volume loop
Dynamic hyperinflation | up to 2 hours during the intervention (exercise)
  Units: % of total lung capacity, measured as change in end-expiratory lung volume from rest to exercise
Forced expiratory volume in 1 s | Pre to 30 min post exercise
  Units: Litres, measured with spirometry
Peripheral airway reactivity (R5-R20) | Pre to 30 min post exercise
  Units: % change from pre to post exercise, measured with impulse oscillometry

SECONDARY OUTCOMES:
Rating of perceived breathlessness | up to 2 hours during the intervention (exercise)
  Borg 0 - 10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Dharini M Bhammar, MBBS, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share all of the individual participant data collected during the trial.